CLINICAL TRIAL: NCT04797026
Title: Reducing Loneliness With Penpal Connections
Brief Title: Penpal Loneliness Project
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to difficulties enrolling given skilled nursing facility staff shortages
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Susan B. Laabs, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-009976
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Loneliness

STUDY DESIGN:
Intervention Model Description: 5 care facility residents paired with a similar amount of students as a pilot. If this program is successful, we will plan to amend IRB to include larger numbers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penpal Program to Alleviate Loneliness (Experimental): A social program connecting patients in residential care facilities with high school students through monthly letter writing would positively impact quality of life for both, reducing quantitative and qualitative measures of loneliness
  Interventions: Other: Letters to increase social connection with goal to alleviate loneliness

INTERVENTIONS:
Other: Letters to increase social connection with goal to alleviate loneliness — Our hypothesis is that a social program connecting patients in residential care facilities with high school students through monthly letter writing would positively impact quality of life for both, reducing quantitative and qualitiative measures of loneliness
  Other Names: Letters

SUMMARY:
The purpose of this research is to study whether sending letters helps reduce loneliness for either the facility resident or the teenager.

DETAILED DESCRIPTION:
Hypothesis: Our hypothesis is that a social program connecting patients in residential care facilities with high school students through monthly letter writing would positively impact quality of life for both, reducing quantitative and qualitiative measures of loneliness

Aims, purpose, or objectives:

Our objective is to reduce loneliness and increase quality of life for patients residing in residential care facilities and for high school students.

Background (Include relevant experience, gaps in current knowledge, preliminary data, etc.):

In response to the Covid pandemic, to protect their residents, residential care facilities have implemented restrictions limiting visitors as well as social activities. Anecdoctally this has negative impacted the quality of life of those residents, increasing their loneliness. Previous studies have shown positive impact of intergenerational programs including penpal programs.

ELIGIBILITY:
Inclusion Criteria:

* Care facility residents with capacity to make decisions:
* Measured via their most recent cognitive assessment;
* Subjectively measured via nursing staff.
* High school students will be invited via recommendation of their instructors and school administrative staff:
* Parental permission will be required.

Exclusion Criteria:

* Care facility residents that have significant cognitive impairment.
* Residents who lack decision-making capacity.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
Loneliness Alleviation with Letter Writing | 6 months; may be extended
  Writing letters between Long Term Care Residents and Students: Increasing Connection to Alleviate Loneliness

CONTACTS AND LOCATIONS:
Overall Officials: Susan Laabs, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials